CLINICAL TRIAL: NCT06607900
Title: A Multi-center, Open, Single-arm, Basket-design Clinical Trial to Evaluate the Safety and Efficacy of Human Umbilical Cord Mesenchymal Stem Cell-derived Small Extracellular Vesicles hUC-MSC-sEV-001 Nasal Drops for the Treatment of Multiple Neurodegenerative Diseases
Brief Title: hUC-MSC-sEV-001 Nasal Drops for Neurodegenerative Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMEC-2024-002
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Parkinson Disease; Lewy Body Dementia; Multiple System Atrophy; Fronto-temporal Dementia; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Lewy Body Disease; Multiple System Atrophy; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hUC-MSC-sEV-001 group (Experimental): hUC-MSC-sEV-001 nasal drops treatment
  Interventions: Drug: hUC-MSC-sEV-001 nasal drops

INTERVENTIONS:
Drug: hUC-MSC-sEV-001 nasal drops — hUC-MSC-sEV-001 nasal drops

SUMMARY:
To evaluate the safety and preliminary efficacy of human umbilical cord mesenchymal stem cell-derived small extracellular vesicles hUC-MSC-sEV-001 nasal drops in multiple neurodegenerative diseases, including Alzheimer's disease, Parkinson's disease, multiple system atrophy, Lewy body dementia, frontotemporal dementia, and amyotrophic lateral sclerosis.

ELIGIBILITY:
General Criteria:

Inclusion Criteria:

1. Age 18-80 years (inclusive), any gender.
2. Subjects or their legal guardians voluntarily sign a written informed consent form and are able to comply with the study requirements for dosing and follow-up.

Exclusion Criteria:

1. Subjects who have received allogeneic mesenchymal progenitor cell therapy or its derived small extracellular vesicles.
2. Subjects with abnormal nasal anatomy, nasal damage, severe rhinitis, or other nasal conditions that may affect the administration of the investigational product.
3. Subjects requiring nasogastric tube insertion.
4. Suffering from other uncontrolled diseases that may interfere with the study results, including but not limited to severe local infection, systemic infection, or immunodeficiency.
5. Combined with malignant tumors, hematological malignancies, or other serious systemic diseases.
6. Clinically significant history of allergic reactions, especially drug allergic reactions.
7. Severe renal insufficiency: creatinine clearance (CrCl) < 30 mL/min (calculated by Cockcroft-Gault formula), or other known severe renal diseases.
8. Peripheral blood hemoglobin (HGB) < 100 g/L, absolute neutrophil count (NEUT) < 1.5 × 10⁹/L, platelet count (PLT) < 100 × 10⁹/L, white blood cell count (WBC) < 4.0 × 10⁹/L or ≥ 12 × 10⁹/L, serum albumin < 30 g/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 × upper limit of normal (ULN).
9. HBsAg positive, or HBcAb positive with HBV DNA positive, hepatitis C virus (HCV) antibody positive, peripheral blood HCV RNA positive, HIV antibody positive; CMV DNA positive, syphilis serology positive.
10. Contraindications to MRI examination (e.g., metal implants) or inability to tolerate MRI (e.g., claustrophobia).
11. Women of childbearing potential not intending to use effective contraception during the trial or within 90 days after the last dose and with a positive pregnancy test record; pregnant or lactating women; men who are sexually active during the trial or within 90 days after the last dose and not intending to use effective contraception; or men planning to donate sperm during the trial or within 90 days after the last dose.
12. Vaccination within 1 month prior to the first dose or planned during the period from enrollment until the end of follow-up.
13. Participation in other clinical drug studies within the past 30 days.
14. Any condition that, in the investigator's judgment, may compromise the subject's ability to understand and/or comply with the study procedures and/or follow-up.

Alzheimer's Disease (AD) Specific Criteria:

Inclusion Criteria:

1. Probable AD as defined by the 2011 National Institute on Aging-Alzheimer's Association (NIA-AA) criteria.
2. Clinical Dementia Rating (CDR) score ≤ 1.0.
3. Subjects have an identified, reliable caregiver.
4. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Major history of significant brain injury with persistent neurological impairment (with or without) or known structural brain abnormalities.
2. Cognitive impairment due to other causes: central nervous system infection, Creutzfeldt-Jakob disease, traumatic dementia, other physical/chemical factors (e.g., drug intoxication, alcoholism, carbon monoxide poisoning), major systemic illnesses (e.g., hepatic encephalopathy, pulmonary encephalopathy), intracranial space-occupying lesions (e.g., subdural hematoma, brain tumor), endocrine disorders (e.g., thyroid disease, parathyroid disease), vitamin B12 or folate deficiency, or any other known causes.

Parkinson's Disease (PD) Specific Criteria:

Inclusion Criteria:

1. Diagnosis of PD according to the 2015 Movement Disorder Society (MDS) clinical diagnostic criteria for PD.
2. Hoehn and Yahr stage ≤ 3.
3. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Parkinsonism other than PD, including but not limited to progressive supranuclear palsy (PSP), multiple system atrophy (MSA), vascular parkinsonism, drug-induced parkinsonism, essential tremor, primary dystonia.

Multiple System Atrophy (MSA) Specific Criteria:

Inclusion Criteria:

1. Diagnosis of possible or probable multiple system atrophy.
2. Time since diagnosis < 3 years from baseline, with an expected survival of at least 3 years.
3. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Modified Unified Multiple System Atrophy Rating Scale (UMSARS) Part I score ≥ 14.
2. Presence of any condition that, in the investigators' judgment, affects the diagnosis or assessment of MSA.

Dementia with Lewy Bodies (DLB) Specific Criteria:

Inclusion Criteria:

1. Meets the revised consensus criteria for DLB (Fourth Consensus Report of the DLB Consortium, 2017).
2. Severity of motor symptoms must be ≤ stage 3 on the Hoehn and Yahr scale.
3. Clinical Dementia Rating (CDR) score ≤ 1.0.
4. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Patients currently diagnosed with any primary psychiatric disorder (e.g., schizophrenia, bipolar disorder, or major depressive episode) according to DSM-V.
2. Patients with clinically significant or unstable systemic illness and exposure to toxicants within the past 5 years.

Frontotemporal Dementia (FTD) Specific Criteria:

Inclusion Criteria:

1. Meets the 2017 International Research Society (IRS) diagnostic criteria for FTD.
2. Clinical Dementia Rating (CDR) score ≤ 1.0.
3. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Diagnosis of severe central nervous system diseases other than FTD that may be the cause of the patient's FTD symptoms or may affect the study objectives.

Amyotrophic Lateral Sclerosis (ALS) Specific Criteria:

Inclusion Criteria:

1. Diagnosis of Amyotrophic Lateral Sclerosis (ALS) meeting the diagnostic criteria (Revised El Escorial Criteria, 2000 or Airlie House Criteria) at the level of definite, probable, or laboratory-supported probable ALS.
2. Disease duration ≥ 6 months and ≤ 2 years (from the first occurrence of any ALS symptom).
3. Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) score: each individual item score ≥ 2 points (with the three respiratory items - Dyspnea, Orthopnea, and Respiratory Insufficiency - all scoring 4 points).
4. Stable treatment regimen for at least 1 month prior to dosing.

Exclusion Criteria:

1. Diagnosis of non-ALS patients based on clinical presentation and available auxiliary clinical examinations (neurophysiology, MRI or other imaging techniques, laboratory tests, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's disease: Change in Alzheimer's disease assessment scale-cognitive section（ADAS-cog） | 12 months
  ADAS-Cog is comprised of 11 modalities that evaluate memory, praxis, and language deficiencies. The total score range is 0 to 70 points, with higher scores indicating greater cognitive impairment.
Parkinson's disease: Change in MDS Unified-Parkinson Disease Rating Scale(MDS-UPDRS) | 12 months
  The MDS-UPDRS is defined by 4 Parts, each composed by a different number of items. The MDS-UPDRS has a minimum score of 0 and a maximum score of 260. The higher the score, the more severe the impairment.
multiple system atrophy: Unified Multiple System Atrophy Rating Scale（Part I and Part II） | 12 months
  UMSARS is a clinical tool designed to assess the severity and progression of MSA. The scale is divided into multiple parts, with Part I focusing on functional disability based on the history and self-report symptoms and Part II the severity of motor symptoms through a physical examination. The higher score, the severer impairment.
lewy body dementia: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) | 12 months
  ADCS-CGIC provides a clinician-rated, subjective evaluation of a patient's cognitive, behavioral, and functional performance based on interviews and observations. The scoring typically uses a 7-point scale. The lower score, the better changes in overall condition.
frontotemporal dementia: CDR Dementia Staging Instrument PLUS National Alzheimer's Coordinating Center Behavior and Language Domains（CDR+NACC FTLD） | 12 months
  The CDR Dementia Staging Instrument provides a global assessment of cognitive and functional decline, while the NACC Behavior and Language Domains offer a more nuanced view of neuropsychiatric symptoms and language impairments.
Amyotrophic lateral sclerosis: Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 6 months
  The ALSFRS-R is rating scale (ratings 0 = can't do, to 4 = normal ability) used to determine participants' assessment of their capability and independence in 12 functional activities.
  This is a validated scale, both in person and by phone, which provides a total score from four sub-scores which assess speech and swallowing (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function).
  Total scores range from 0 (most impaired) to 48 (normal ability).

SECONDARY OUTCOMES:
Barthel index | 6 months, 12months
  The Barthel Index is used for measuring a person&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s ability to perform basic activities of daily living.Scores typically range from 0 (totally dependent) to 100 (completely independent), with higher scores indicating greater independence in daily functioning.
mini mental status exam(MMSE) | 6 months, 12months
  The Mini-Mental State Examination (MMSE) is used for assessing cognitive function. The MMSE is scored out of a total of 30 points. A higher score indicates better cognitive function.
EQ-5D-5L | 6 months, 12months
  The EQ-5D-5L is used to measure health-related quality of life. The EQ-5D-5L assesses health on a scale of 0 to 25. A higher score means a lower quality of life.
Alzheimer's disease: sum of boxes of the CDR（CDR-SB） | 6 months, 12months
  The CDR-SB is used to assess the severity of cognitive impairment and dementia. The total score can range from 0 to 18, where higher scores indicate greater levels of impairment across the domains.
Alzheimer's disease: Alzheimer's Disease Cooperative Study - Activities of Daily Living （ADCS-ADL） | 6 months, 12months
  The ADCS-ADL is used to assess functional decline in patients with Alzheimer's disease, especially in the mild to moderate stages. The total score ranges from 0 to 78 , with higher scores indicating greater functional independence.
multiple system atrophy: Composite Autonomic Symptom Score | 6 months, 12months
  The COMPASS questionnaire is used to evaluate autonomic dysfunction, which can present with a variety of symptoms.Higher scores indicate greater impairment in autonomic function.
Clinical Global Impression | 6 months, 12months
  CGI is used to assess the severity of a patient's illness, the change in their condition over time, and the efficacy of treatments. It is scored on a 7-point scale, with a higher score indicating a worsen condition.
lewy body dementia: MDS-UPRDS | 6 months, 12months
Lewy body dementia：Neuropsychiatric Inventory（NPI） | 6 months, 12months
  NPI is used to assess neuropsychiatric symptoms and behavioral disturbances in individuals. The Total NPI Score ranges from 0 to 144. Higher scores indicate greater overall severity of neuropsychiatric disturbances.
frontotemporal dementia: NPI | 6 months, 12months
frontotemporal dementia: ADAS-cog | 6 months, 12months
Amyotrophic lateral sclerosis: Change in forced vital capacity to predicted value ratio (FVC% pred) | 6 months
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration.
Amyotrophic lateral sclerosis: Change in the Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40). | 6 months
  ALSAQ-40 score ranges from 0 to 160 points, and higher scores indicate better quality of life.
Amyotrophic lateral sclerosis: Change in the Edinburgh Cognitive and Behavioral ALS Screen (ECAS). | 6 months
  ECAS determine cognitive and behavioral changes of patients suffering from Amyotrophic Lateral Sclerosis.
  With ECAS, ALS-specific (fluency, executive functions and social cognition, language; minimum score = 0, maximum score = 100) and ALS-nonspecific (memory, visuospatial functions; minimum score = 0, maximum score = 36) functions can be analyzed to enable the distinction from other diseases with cognitive and behavioral impairments.
Amyotrophic lateral sclerosis: Change in the Neurophysiological Index (NI) and Compound Muscle Action Potential (CMAP) score. | 6 months
  The NI is derived from the CMAP, the DML and the F-wave frequency (CMAP amplitude/DML) x F frequency %), representing aspects of the effects of denervation and reinnervation, of degeneration of the terminal part of the motor axons, and of the excitability of anterior horn cells.
  The negative amplitudes of the CMAP for motor nerve conduction in the median and ulnar nerves in the upper extremities as well as the peroneal and tibial nerves in the lower extremities of ALS patients were recorded (median nerve-wrist, ulnar-wrist, peroneal-ankle, tibial-ankle). These nerves were scored based on the decrease in the amplitudes of each nerve CMAP- 0 (CMAP> =[X-2s]), 1 (50% [X-2s] < CMAP < [X-2s]), 2 (30% [X-2s] < CMAP < 50% [X-2s]), 3 (CMAP < =30% [X-2s]), respectively. The values of X and S for different nerves and different patient age groups, which were applied in the electrophysiology examination room.
Amyotrophic lateral sclersis: Change in the Rasch Overall ALS Disability Scale (ROADS). | 6 months
  ROADS score ranges from 0 to 56 points, and higher scores indicate better basic daily function.
Adverse effects | 3months, 6 months, 12months

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided